Study Title: 4DCT Wrist Biomarkers During Resisted and Unresisted Tasks in Healthy Controls

Document Date: 16 November 2022

NCT#: NCT04736537



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

# RESEARCH PARTICIPANT CONSENT AND PRIVACY AUTHORIZATION FORM

**Study Title:** 4DCT Wrist Biomarkers during Resisted and Unresisted Tasks in Healthy

Controls

**IRB#:** 20-007668

Principal Investigator: Kristin Zhao, Ph.D., and Colleagues

# **Key Study Information**

This section provides a brief summary of the study. It is important for you to understand why the research is being done and what it will involve before you decide. Please take the time to read the entire consent form carefully and talk to a member of the research team before making your decision. You should not sign this form if you have any questions that have not been answered. This is a research study. Being in this research study is your choice; you do not have to participate. If you decide to join, you can still stop It's Your Choice at any time. You should only participate if you want to do so. You will not lose any services, benefits or rights you would normally have if you choose not to take part. The purpose of this research is to examine gapping in wrist joint bones during wrist movement, and to determine whether, and how much, the size of these gaps changes if light resistance is applied to the **Research Purpose** movements. You are being asked to take part in this research study because you have no known history of wrist-related injury or disease. What's Involved Study participation involves a single visit to have computerized tomography (CT) scans of your forearms. You will be exposed to radiation from the CT scans. The amount of **Key Information** radiation has a low risk of harmful effects.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

| | If you are interested in learning more about this study, read the rest of this form carefully. The information in this form will help you decide |
|---|---|
| Learn More | if you want to participate in this research or not. A member of our |
| | research team will talk with you about taking part in this study before |
| | you sign this form. If you have questions at any time, please ask us. |

# **Making Your Decision**

Taking part in research is your decision. Take your time to decide. Feel free to discuss the study with your family, friends, and healthcare provider before you make your decision. Taking part in this study is completely voluntary and you do not have to participate.

If you decide to take part in this research study, you will sign this consent form to show that you want to take part. We will give you either a printed or electronic copy of this form to keep. A copy of this form will be put in your medical record.

For purposes of this form, Mayo Clinic refers to Mayo Clinic in Arizona, Florida and Rochester, Minnesota; Mayo Clinic Health System; and all owned and affiliated clinics, hospitals, and entities.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023 Name and Clinic Number

# **Contact Information**

| If you have questions about | You can contact |
|---|---|
| <ul> <li>Study tests and procedures</li> <li>Materials you receive</li> <li>Research-related appointments</li> </ul> | Principal Investigator: Kristin Zhao, Ph.D. Phone: (507) 284-8942 |
| <ul> <li>Research-related concern or complaint</li> </ul> | Study Team Contact: Tyson Scrabeck |
| <ul><li>Research-related injuries or emergencies</li><li>Withdrawing from the research study</li></ul> | <b>Phone:</b> (507) 538-1016 |
| · · | Institution Name and Address: |
| | Mayo Clinic |
| | 200 1 <sup>st</sup> St. SW |
| | Rochester, MN 55905 |
| ■ Rights of a research participant | Mayo Clinic Institutional Review Board (IRB) Phone: (507) 266-4000 Toll-Free: (866) 273-4681 |
| <ul> <li>Rights of a research participant</li> <li>Any research-related concern or complaint</li> <li>Use of your Protected Health Information</li> <li>Stopping your authorization to use your Protected Health Information</li> </ul> | Research Participant Advocate (RPA)<br>(The RPA is independent of the Study Team)<br>Phone: (507) 266-9372<br>Toll-Free: (866) 273-4681 |
| <ul> <li>Withdrawing from the research study</li> </ul> | E-mail: researchparticipantadvocate@mayo.edu |
| <ul> <li>Billing or insurance related to this research</li> </ul> | Patient Account Services |
| study | <b>Toll-Free:</b> (844) 217-9591 |

#### Other Information:

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

A description of this research study will be available on <a href="http://www.mayo.edu/research/clinical-trials">http://www.mayo.edu/research/clinical-trials</a>. This website will not include information that can identify you. You can search this website at any time.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

# Why are you being asked to take part in this research study?

You are being asked to take part in this research study because you have no known history of wrist-related injury or disease.

# Why is this research study being done?

The purpose of this study is to use Four-Dimensional CT imaging (4DCT) and CT motion pictures to visualize and record how much space there is between certain wrist joint bones, both without any resistance, and with light resistance to the movement.

# Information you should know

#### Who is Funding the Study?

The National Institutes of Health (NIH) is funding the study. The NIH will pay the institution to cover costs related to running the study.

# How long will you be in this research study?

You will be in this study for a single CT scanning session (approximately 30 minutes).

# What will happen to you while you are in this research study?

If you agree to be in the study, you will be asked to participate in the following:

This study involves one visit to have five computerized tomography (CT) scans of your joint, without any iodine contrast injection. Four-dimensional CT imaging is the same as a standard



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

CT; however, we are able to image your joint while it is moving instead of in one fixed position. One of the CT scanners which may be used is an experimental device with additional capabilities; this device has not been approved for general use by the Food and Drug Administration (FDA), but it has been approved for use in this study by Mayo Clinic's Institutional Review Board.

The CT scan appointment should take approximately 30 minutes.

The CT Technician will ask you to lay face-down on a table with your arms extended in front of you (i.e. the "Superman" pose). The table moves through a big donut-shaped machine that will then take CT scans (x-rays) of your lower arms, wrists, and hands. Your forearms will be restrained in a padded support channel to help keep arm and shoulder motion from affecting wrist and hand movement. You will be instructed by the CT technician to move your joints during the CT scan, in rhythm to a metronome. For two of the moving scans, a hand-grip device which provides light resistance to flexing and rotating your wrists will be used. The CT scan will take several seconds to complete. You will have a total of five CT scans: one from hand to elbow performed while holding both your hands and arms still; and four of your wrists while moving as instructed (two scans on each arm independently).

Tests done only for research purposes are not meant to provide clinical information or help care for you. The results are only important for research. Therefore, the results of tests done with your information and samples will not be provided to you. In the rare event that a finding might affect the health of you or your family, we will contact you and you can choose whether to receive or refuse the information. If you decide to follow up and further medical testing or care is needed, the costs will be billed to you or your insurance.

# What are the possible risks or discomforts from being in this research study?

You will be exposed to x-ray radiation during the CT scans of your joint. The amount of radiation you will receive has a low risk of harmful effects.

As with all research, there is a chance that confidentiality could be compromised; however, we take precautions to minimize this risk.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

# Are there reasons you might leave this research study early?

You may decide to stop at any time. In addition, the Principal Investigator or Mayo Clinic may stop you from taking part in this study at any time:

- If it is in your best interest,
- If you don't follow the study procedures,
- If the study is stopped.

If you leave this research study early, or are withdrawn from the study, no more information about you will be collected; however, information already collected about you in the study may continue to be used.

# What if you are injured from your participation in this research study?

#### Where to get help:

If you think you have suffered a research-related injury, you should promptly notify the Principal Investigator listed in the Contact Information at the beginning of this form. Mayo Clinic will offer care for research-related injuries, including first aid, emergency treatment and follow-up care as needed.

#### Who will pay for the treatment of research related injuries?

Care for such research-related injuries will be billed in the ordinary manner, to you or your insurance. Treatment costs for research-related injuries not covered by your insurance will be paid by Mayo Clinic.

# What are the possible benefits from being in this research study?

You won't benefit from taking part in this research study. It is for the benefit of research.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

# What alternative do you have if you choose not to participate in this research study?

This study is only being done to gather information. You may choose not to take part in this study.

# What tests or procedures will you need to pay for if you take part in this research study?

You won't need to pay for tests and procedures which are done just for this research study. These tests and procedures are:

CT scans

However, you and/or your insurance will need to pay for all other tests and procedures that you would have as part of your clinical care, including co-payments and deductibles.

If you have billing or insurance questions call Patient Account Services at the telephone number provided in the Contact Information section of this form.

# Will you be paid for taking part in this research study?

You will receive \$50.00 for completing the study visit.

Payment for participation in research is considered taxable income and reportable to the Internal Revenue Service (IRS). Accounts Payable at Mayo Clinic will be given your name, address and Social Security number in order to issue a check for your study participation. If you receive research payments totaling \$600 or more in a calendar year, a tax Form 1099 will be sent to you. For Mayo Clinic employees, research payments are included in your paycheck with applicable taxes withheld and reported on your Form W2 after calendar year-end.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

# Will your information or samples be used for future research?

Identifiable information such as your name, Mayo Clinic number, or date of birth may be removed from your information or samples collected in this study, allowing the information or samples to be used for future research or shared with other researchers without your additional informed consent.

#### How will your privacy and the confidentiality of your records be protected?

Mayo Clinic is committed to protecting the confidentiality of information obtained about you in connection with this research study.

Study data will be kept on secured servers, password-protected computers and file storage devices, and in the researchers' limited-access workspaces.

During this research, information about your health will be collected. Under Federal law called the Privacy Rule, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use and share your health information for research and why they may need to do so. Information about you and your health cannot be used in this research study without your written permission. If you sign this form, it will provide that permission (or "authorization") to Mayo Clinic.

# Your health information may be collected from:

- Past, present and future medical records.
- Research procedures, including research office visits, tests, interviews and questionnaires.

# Your health information will be used and/or given to others to:

- Do the research.
- Report the results.
- See if the research was conducted following the approved study plan, and applicable rules and regulations.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

# Your health information may be used and shared with:

- Mayo Clinic research staff involved in this study.
- Other Mayo Clinic staff involved in your clinical care.
- The Mayo Clinic Institutional Review Board that oversees the research.
- Federal and State agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health and other United States agencies) or government agencies in other countries that oversee or review research.

### How your information may be shared with others:

While taking part in this study, you will be assigned a code that is unique to you, but does not include information that directly identifies you. This code will be used if your study information is sent outside of Mayo Clinic. The groups or individuals who receive your coded information will use it only for the purposes described in this consent form.

If the results of this study are made public (for example, through scientific meetings, reports or media), information that identifies you will not be used.

In addition, individuals involved in study oversight and <u>not</u> employed by Mayo Clinic may be allowed to review your health information included in past, present, and future medical and/or research records. This review may be done on-site at Mayo Clinic or remotely (from an off-site location). These records contain information that directly identifies you. However, the individuals will not be allowed to record, print, or copy (using paper, digital, photographic or other methods), or remove your identifying information from Mayo Clinic.

# Is your health information protected after it has been shared with others?

Mayo Clinic asks anyone who receives your health information from us to protect your privacy; however, once your information is shared outside Mayo Clinic, we cannot promise that it will remain private and it may no longer be protected by the Privacy Rule.

# **Your Rights and Permissions**

Participation in this study is completely voluntary. You have the right not to participate at all. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to sign this form, but if you do not, you cannot take part in this research study.

Deciding not to participate or choosing to leave the study will not result in any penalty. Saying 'no' will not harm your relationship with your own doctors or with Mayo Clinic.

IRB#: 20-007668 00 Page 9 of 11 IRB Doc. Ctrl # 10013.34



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

If you cancel your permission for Mayo Clinic to use or share your health information, your participation in this study will end and no more information about you will be collected; however, information already collected about you in the study may continue to be used.

You can cancel your permission for Mayo Clinic to use or share your health information at any time by sending a letter to the address below:

Mayo Clinic
Office for Human Research Protection
ATTN: Notice of Revocation of Authorization
201 Building 4-60
200 1st Street SW
Rochester, MN 55905

Alternatively, you may cancel your permission by emailing the Mayo Clinic Research Participant Advocate at: <a href="mailto:researchparticipantadvocate@mayo.edu">researchparticipantadvocate@mayo.edu</a>.

Please be sure to include in your letter or email:

- The name of the Principal Investigator,
- The study IRB number and /or study name, and
- Your contact information.

Your permission for Mayo Clinic to use and share your health information lasts until the end of this study, unless you cancel it. The study does not end until all data has been collected, checked (or audited), analyzed, and reported. Because research is an ongoing process, we cannot give you an exact date when the study will end. Sometimes this can be years after your study visits and/or activities have ended.



Approval Date: November 16, 2022 Not to be used after: November 3, 2023

| Enrollment and Permission Signatures | | | |
|---|---|---|---|
| Your signature documents your permission to take part in this research. | | | |
| | / / Date | : | AM/PM |
| Printed Name | Date | Time | |
| Signature | | | |
| Person Obtaining Consent • I have explained the t | research study to the participant. | | |
| | uestions about this research study t | o the best of my abili | ty. |
| | / / | : | AM/PM |
| Printed Name | Date | Time | |
| Signature | | | |